CLINICAL TRIAL: NCT00396864
Title: Phase 1 Clinical Trial of NPI-0052 in Patients With Advanced Solid Tumor Malignancies or Refractory Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPI-0052-100; NCT00385814 (obsolete NCT alias)
Record Dates: First submitted 2006-11-06; First posted 2006-11-08 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Cancer; Lymphomas
Keywords: cutaneous lymphoma; marginal zone lymphoma
MeSH Terms: conditions — Neoplasms; Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, B-Cell, Marginal Zone | interventions — marizomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NPI-0052 (Experimental): Advanced Solid Tumor Malignancies and Refractory Lymphoma
  Interventions: Drug: NPI-0052

INTERVENTIONS:
Drug: NPI-0052 — NPI-0052 IV injection at doses ranging from 0.0125 to 0.8 mg/m2 over 1 to 10 minutes on Day 1, Day 8, Day 15 of each 28-day Cycle; 11 dose cohorts during dose-escalation
  Other Names: Marizomib; MRZ

SUMMARY:
Multicenter, open-label study of NPI-0052 in patients with advanced solid tumor malignancies or refractory lymphoma whose disease had progressed after treatment with standard, approved therapies that included 2 stages. The initial stage involved dose escalation to an MTD and determination of a recommended Phase 2 dose. The second stage comprised an expansion cohort at the recommended Phase 2 dose.

DETAILED DESCRIPTION:
NPI-0052 (also known as marizomab) is a second generation proteasome inhibitor being developed as an anticancer agent. Proteasomes are responsible for degrading substrates such as damaged and aged proteins, tumor suppressors, and cell cycle regulators, and for regulating NF-κB activation by degrading its inhibitor, IκB. Blocking the proteasome pathway results in accumulation of proteins, which can cause cell death, particularly in tumor cells (Kisselev, 2001).

The Food and Drug Administration (FDA) approved the first proteasome inhibitor (bortezomib; Velcade®) in 2003 for the treatment of patients with multiple myeloma (MM) and subsequently for treatment of patients with mantle cell lymphoma in 2006. Although this compound has demonstrated efficacy in both of those indications, resistance and toxicity develop with continued therapy. Resistance may result from a variety of mechanisms. Bortezomib toxicity (primarily neurological with peripheral neuropathy and neuralgia, and also thrombocytopenia and neutropenia) can result in treatment discontinuation (about 25% of patients in a clinical trial conducted in patients at time of first relapse required cessation of therapy due to adverse events).

NPI-0052 inhibits the chymotrypsin-like (CT-L), caspase-like (C-L), and trypsin-like (T-L) activity of human erythrocyte-derived 20S proteasomes. Also known as salinosporamide A, NPI-0052 is a novel chemical entity discovered during the fermentation of Salinispora tropica NPS021184, a marine actinomycete, and is manufactured by saline fermentation. NPI-0052 was shown in nonclinical studies to have increased potency and duration of biological effects compared with bortezomib and may provide a significant therapeutic advantage, particularly if toxicity is less at therapeutic doses.

This was the first-in-human study of NPI-0052, and was conducted in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed solid tumor malignancy (patients must be refractory to or demonstrate unacceptable toxicity towards effective therapy known to provide clinical benefit for their condition) OR refractory lymphoma (patients whose disease has progressed despite standard therapy including at least one-doxorubicin-containing regimen and one anti-CD20 monoclonal antibody-containing regimen.
* KPS ≥70%.
* All Adverse Events of any prior chemotherapy, surgery, or radiotherapy, must have resolved to NCI CTCAE (v. 3.0) Grade ≤ 1 (except for hemoglobin).
* Adequate bone marrow, renal, adrenal, pancreatic and liver function.
* Signed informed consent.

Exclusion Criteria:

* Administration of chemotherapy, biological, immunotherapy or investigational agent (therapeutic or diagnostic) within 28 days prior to receipt of study medication (6 weeks for nitrosoureas or mitomycin C; 12 weeks for radioimmunotherapy). Major surgery, other than diagnostic surgery, within 4 weeks before first study drug administration. Radiotherapy within 4 weeks.
* Patients that require G-CSF and/or platelet support.
* Patients with ongoing coagulopathies.
* Patients with prior bone marrow transplant therapy (autologous or allogeneic).
* Patients receiving intrathecal therapy.
* Known brain metastases.
* Significant cardiac disease.
* Patients with a prior hypersensitivity reaction of CTCAE Grade ≥ 3 to therapy containing propylene glycol or ethanol.
* Pregnant or breast-feeding women. Female patients must be postmenopausal, surgically sterile or they must agree to use acceptable methods of birth control. Female patients with childbearing potential must have a negative serum pregnancy test. Male patients must be surgically sterile or agree to use an acceptable method of contraception.
* Concurrent, active secondary malignancy for which the patient is receiving therapy.
* Active uncontrolled bacterial or fungal infection requiring systemic therapy; infection requiring parenteral antibiotics.
* Known to be positive for HIV; active hepatitis A, B, or C infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety | Continuous
Maximum Tolerated Dose (MTD) | Continuous
Pharmacokinetics | Continuous

SECONDARY OUTCOMES:
Pharmacodynamics | Continuous
Response | Continous

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Reich, MD, Study Director — Triphase Research and Development I Corp
Locations (3):
- United States (3):
  - Premiere Oncology of America, Scottsdale, Arizona
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Univ. of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided